CLINICAL TRIAL: NCT06273046
Title: Tratamiento de la Incontinencia Fecal y Los Trastornos Funcionales de la defecación Mediante Biofeedback no Instrumental
Brief Title: Treatment of Fecal Incontinence and Functional Evacuation Disorders Using Non-instrumental Biofeedback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)614/2023
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-07-06 (Actual); Status verified 2025-07

CONDITIONS: Fecal Incontinence; Outlet Dysfunction Constipation
MeSH Terms: conditions — Fecal Incontinence | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biofeedback (Experimental)
  Interventions: Behavioral: Biofeedback
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Biofeedback — Three visits will be made throughout the study. The first visit (Day -14) will consist of an evaluation of the inclusion criteria. A pre-treatment anorectal manometry will be performed, and a daily symptom questionnaire will be given to the patient. The second visit will take place 14 days later (Day 0). During this visit, the daily clinical symptom questionnaire will be collected and it will be verified that the patient meets the inclusion criteria. Patients who meet the criteria will be randomized 2:1 to active treatment or placebo. Patients will receive instructions, by means of psychoeducational videos on the exercises to be performed daily at home. A final visit will be performed at the end of the study (3 months in incontinence studies and 4 weeks in dyssynergic defecation studies). In incontinence study a final phone call will be performed at 6 months.
  Arms: Biofeedback
Behavioral: Placebo — Three visits will be made throughout the study following the same procedure as patients in the active arm. Patients randomized to placebo treatment will receive instructions to take a pill of placebo containing 0.3 g glucose daily at home. A final visit will be performed at the end of the study alike the active treatment group.
  Arms: Placebo

SUMMARY:
Background. Rehabilitation and re-education using instrumental anorectal biofeedback are the main treatment of anorectal functional disorders producing incontinence and outlet obstructed defecation. These treatments imply intubation of patient and several sessions of treatment leading to high consumption of resources and costs.

Hypothesis. A cognitive intervention based on original audiovisual programs developed specifically for the management of anorectal functional disorders is effective in correcting anorectal function disorders that cause fecal incontinence and evacuation disorders.

Aim. To prove in two different protocols (fecal incontinence and dyssinergic defecation) the efficacy of specifically developed non-instrumental biofeedback techniques.

Selection criteria. Patients with fecal incontinence and altered sphincter function and patients with outlet obstructed evacuation referred for biofeedback treatment.

Intervention. In separate studies (incontinence and dyssynergic defecation) patients will be randomized into biofeedback and placebo groups. One session of either biofeedback or placebo intervention will be performed at the beginning of the intervention period and patients will be instructed to performed the assigned daily treatment at home. A visit for outcome assessment will be performed at 3 months in incontinence study and at 4 weeks in the dyssinergic defecation study. In addition, in the incontinence study a phone call will be performed after 6 months of the beginning of the study to evaluate treatment outcome.

Biofeedback: patients will be taught to control anal and abdominal muscular activity by providing instructions using original video supports. Patients will be instructed to perform the same exercises daily at home in scheduled times.

Placebo: a pill of placebo containing 0.3 g glucose will be administered every day at home.

ELIGIBILITY:
Inclusion Criteria:

Incontinence studies

* Patients who have at least 4 episodes of fecal incontinence during the last 14 days.
* Patients able to follow instructions and attend study visits.

Dyssinergic defecation studies

* Patients with constipation who present less than 3 complete spontaneous bowel movements per week and/or who have Bristol 1 or Bristol 2 type stools in more than 25% of the bowel movements in the 2 weeks prior to the study
* Patients able to follow instructions and attend study visits.

Exclusion Criteria:

* Patients with organic digestive diseases such as inflammatory bowel disease, celiac disease, gastro-duodenal ulcer...
* Patients with neurological diseases (spinal cord injury, multiple sclerosis, Parkinson's disease).
* Patients with previous of active colon and/or rectal cancer.
* Patients with rectal fistula.
* Patients with rectal prolapse.
* Patients with total colectomy.
* Patients who have had any radiation to the pelvis in the last month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Fecal incontinence study: Number of anal leaks | 3 months
  Number of involuntary leaks during the last 15 days of study compared to the 15 days prior to treatment start.
Dyssinergic defecation study: Number of bowel movements | 4 weeks
  Number and type (according to Bristol scale) of bowel movements during the last 15 days of study compared to the 15 days prior to treatment start.

SECONDARY OUTCOMES:
Incontinence study: Wexner scale | 3 and 6 months
  Score rated at the end of the study compared to the score rated prior to treatment start using the Wexner scale for incontinence.
Incontinence study: Quality of life | 3 months
  Score rated at the end of the study compared to the score rated prior to treatment start using the quality of life questionnaire for incontinence (FIQoL)
Incontinence study: anxiety and depression | 3 months
  Score rated at the end of the study compared to the score rated prior to treatment start using the hospital anxiety-depression questionnaire (HDA)
Incontinence study: Anal sphincter function | 3 months
  Resting pressure and squeeze pressure of the anal sphincters at the end of the study compared to pressures prior to treatment start measured by anorectal manometry
Dyssinergic defecation study: sensation of outlet obstructed evacuation | 4 weeks
  Frequency of the following sensations: sensation of anorectal obstruction/blockage; straining; incomplete evacuation; manual maneuvers to facilitate evacuation during the bowel movements produced during the last 15 days of study compared to the 15 days prior to treatment start using daily questionnaires.
Dyssinergic defecation study: Wexner scale | 4 weeks
  Score rated at the end of the study compared to the score rated prior to treatment start using the Wexner scale for constipation
Dyssinergic defecation study: Quality of life | 4 weeks
  Score rated at the end of the study compared to the score rated prior to treatment start using the patient assessment quality of life questionnaire for constipation (PACQoL)
Dyssinergic defecation study: anxiety and depression | 4 weeks
  Score rated at the end of the study compared to the score rated prior to treatment start using the hospital anxiety-depression questionnaire (HDA)
Dyssinergic defecation study: defecatory maneuvers | 4 weeks
  Abdominal contraction pressure and anal relaxation of the anal sphincters at the end of the study compared to pressures prior to treatment start measured by anorectal manometry

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Serra, MD, Principal Investigator — University Hospital Vall d'Hebron
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serra J, Pohl D, Azpiroz F, Chiarioni G, Ducrotte P, Gourcerol G, Hungin APS, Layer P, Mendive JM, Pfeifer J, Rogler G, Scott SM, Simren M, Whorwell P; Functional Constipation Guidelines Working Group. European society of neurogastroenterology and motility guidelines on functional constipation in adults. Neurogastroenterol Motil. 2020 Feb;32(2):e13762. doi: 10.1111/nmo.13762. Epub 2019 Nov 22. PMID 31756783